CLINICAL TRIAL: NCT02929342
Title: An Open Label, Single-Period Repeated Dose Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Pitolisant, at Steady-State Conditions, in Healthy CYP2D6 Genotyped Male Subjects
Brief Title: Study to Assess the Absorption, Distribution, Metabolism and Excretion (ADME) of [14C]-Pitolisant in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P15-02 / Pitolisant; 2016-000748-32 (EudraCT Number)
Record Dates: First submitted 2016-10-06; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pitolisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitolisant (Experimental): Pitolisant, oral single dose administration, from Day1 to Day7.
  Interventions: Drug: Pitolisant
- [14C]-Pitolisant (Experimental): [14C]-Pitolisant, oral single dose administration at Day8.
  Interventions: Radiation: [14C]-Pitolisant

INTERVENTIONS:
Drug: Pitolisant
  Arms: Pitolisant
Radiation: [14C]-Pitolisant
  Arms: [14C]-Pitolisant

SUMMARY:
The purpose of this study is to better define the absorption and elimination pathways, and circulating metabolites of Pitolisant at steady state using Pitolisant radiolabelled, in healthy CYP2D6 genotyped male subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 30 to 65 years.
* Body mass index 18.0 to 35.0 kg/m2.
* Genotyped with regard to their CYP2D6 status.

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.
* Regular alcohol consumption in males >21 units per week.
* Current smokers and those who have smoked within the last 12 months.
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the Cockcroft-Gault equation.
* Use of CYP2D6 inhibitors or inducers in the 28 days prior to IMP administration

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity (Ae) in urine, faeces and expired air. | from Day 8 (pre-dose) to 120 h post 14C-radioactivity dose
Peak Plasma Concentration (Cmax), pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose
Area under the plasma concentration versus time curve [AUC(0-tau), AUC(0-inf), %AUCextrap], pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose
Volume of distribution (Vz/F), pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose
Apparent clearance (Clss/F), pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose
The slope of the apparent elimination phase (lambda-z), pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose
The apparent elimination half-life (T½), pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose
Time to reach Cmax (Tmax), pitolisant and major metabolites. | From Day 1 (pre-dose) until 168hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MD, Principal Investigator — Quotient Clinical; Thierry Duvauchelle, MD, Study Director — Bioprojet Pharma